CLINICAL TRIAL: NCT01972477
Title: The Effect of DLBS1449 in Diabetic Patients With Low HDL-Cholesterol - Double Blind Comparative Study With Placebo
Brief Title: DLBS1449 in Diabetic Patients With Low HDL
Status: Withdrawn | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Dexa Medica Group (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DLBS1449-0111
Record Dates: First submitted 2013-10-24; First posted 2013-10-30 (Estimated); Last update posted 2016-08-04 (Estimated); Status verified 2016-08

CONDITIONS: Diabetic Patients; Low HDL-cholesterol (< 35 mg/dL); Lifestyle Intervention for at Least 1 Month
Keywords: DLBS1449; diabetes mellitus; HDL-cholesterol
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- DLBS1449, 1x75 mg (Experimental): DLBS1449 softcapsule 1x75 mg daily, taken every day along the study period.
  Interventions: Drug: DLBS1449
- DLBS1449, 1x150 mg (Experimental): DLBS1449 softcapsule 1x150 mg (2 softcapsules 75 mg) daily, taken every day along the study period
  Interventions: Drug: DLBS1449
- Placebo (Placebo Comparator): Placebo once daily, taken every day along the study period
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: DLBS1449 — Study treatment will be DLBS1449 softcapsules at a dose of 1x75 mg daily or DLBS1449 at a dose of 1x150 mg daily. DLBS1449 will be given every day for 8 weeks.
  Other Names: Forhidrol
  Arms: DLBS1449, 1x150 mg; DLBS1449, 1x75 mg
Other: Placebo — Placebo will be given every day for 8 weeks.
  Arms: Placebo

SUMMARY:
This is a parallel, 3-arm, randomized, prospective, placebo-controlled, and double-blind clinical study for eight weeks of therapy to investigate the clinical efficacy of DLBS1449 in elevating high density lipoprotein (HDL) cholesterol in diabetic patients. The hypothesis of interest for the study is: the administration of DLBS1449 will elevate HDL-cholesterol level from baseline to the end of study significantly higher than the elevation resulted by placebo. In addition, the administration of DLBS1449 at the dose of 150 mg daily will provide a significantly better response than that of the lower dose (DLBS1449 75 mg daily).

DETAILED DESCRIPTION:
There will be three groups of treatment by dosage regimen in this study. Eligible subjects will be randomized to receive any of the following regimens: 1) DLBS1449 at a dose of 1 x 75 mg daily, or 2) DLBS1449 at a dose of 1 x 150 mg (two capsules of DLBS1449 75 mg) daily; or 3) placebo, once daily. Study medication should be administered once daily, in the evening with meal, for eight weeks. Clinical and laboratory examinations to evaluate investigational drug's efficacy and safety will be performed at baseline and at interval of four weeks over 8-week course of therapy.

ELIGIBILITY:
Inclusion Criteria:

* Male or female 21 - 70 years.
* Have been diagnosed diabetes mellitus and being treated with lifestyle intervention for at least 1 month prior to screening, with or without antidiabetic agents.
* HDL-cholesterol level of < 35 mg/dL.
* Triglycerides level of < 200 mg/dL.
* Adequate liver and renal function.
* Statin and/or fenofibrate therapy should have been being regularly taken for >=3 months at stable dose (ONLY for subjects currently under statin and/or fenofibrate therapy).
* Able to take oral medication.

Exclusion Criteria:

* Pregnant or breast-feeding women or willing to be pregnant.
* Symptomatic congestive heart failure, unstable angina pectoris, or cardiac arrhythmia.
* Uncontrolled hypertension (SBP > 160 mmHg and/or DBP > 100 mmHg).
* Any other disease state, including chronic/acute systemic infections, uncontrolled illnesses or other chronic diseases, which judged by the investigator, could interfere with trial participation or trial evaluation.
* Concurrent treatment with systemic corticosteroids or herbal (alternative) medicines.
* Known allergic or hypersensitive to drugs contain similar active substance with the study medication.
* Participation in any other clinical studies within 30 days prior to screening.

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-07; Primary Completion 2017-10 (Estimated); Study Completion 2018-01 (Estimated)

PRIMARY OUTCOMES:
Percent change in HDL-cholesterol level | 8 weeks

SECONDARY OUTCOMES:
Percent change in HDL-cholesterol level | 4 and 8 weeks
Percent change in LDL-cholesterol level | 4 and 8 weeks
Percent change in sd LDL-cholesterol level | 4 and 8 weeks
Percent change in triglycerides level | 4 and 8 weeks
Percent change in total cholesterol level | 4 and 8 weeks
Change in Apo-A1 | 4 and 8 weeks
Change in Apo-B | 4 and 8 weeks
Response rate | 8 weeks
  Response rate is defined as percentage of subjects with HDL-cholesterol >= 40 mg/dL after 8 weeks of treatment.
Change in A1c level | 8 weeks
Vital signs | 4 and 8 weeks
  Vital signs measurements include: blood pressure, heart rate, and respiratory rate.
Routine hematology | 4 and 8 weeks
  Routine hematology measurements include: hemoglobin, hematocrit, RBC, WBC, differentiation of WBC, and platelet count.
Liver function | 4 and 8 weeks
  Liver function measurements include: serum ALT, serum AST, gamma-GT, and alkaline phosphatase.
Renal function | 4 and 8 weeks
  Renal function measurement includes: serum creatinine.
Electrocardiography (ECG) | 8 weeks
  The interpretation of ECG result will be recorded. Any worsened changes from baseline condition will be counted as adverse events.
Adverse event | 1-8 weeks
  Adverse event will be observed and recorded during the study period.

CONTACTS AND LOCATIONS:
Overall Officials: Askandar Tjokroprawiro, Prof, SpPD, K-EMD, FINASIM, MD, Principal Investigator — Surabaya Diabetes and Nutrition Center, Dr. Soetomo Hospital
Locations (1):
- Surabaya Diabetes and Nutrition Center, Dr. Soetomo Hospital; Pusat Diagnostik Terpadu Building 7th Floor, Surabaya, East Java, Indonesia